CLINICAL TRIAL: NCT03207191
Title: A Phase I Study of the Tumor-targeting Human F16IL2 Monoclonal Antibody-cytokine Fusion Protein in Combination With the Anti-CD33 Antibody BI 836858 in Patients With AML Relapse After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Trial to Find and Investigate a Safe Dose of F16IL2 and BI 836858 in Patients With AML Relapse After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: PHIBI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-F16IL2CD33-03/15
Record Dates: First submitted 2016-12-16; First posted 2017-07-02 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Acute Myeloid Leukemia (AML) Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — BI 836858

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- F16IL2 + BI 836858 (Experimental): Successive cohorts of patients will receive increasing doses of FI6IL2 and BI 836858 until the MTD is reached. The MTD will be defined following a Bayesian logistic regression model (BLRM) with overdose control.
  Patients will go off treatment after 6 months (i.e. after 6 cycles of induction combination therapy). Patients achieving CR or CRi will receive maintenance therapy for a maximum of 6 months.
  Interventions: Drug: F16IL2; Drug: BI 836858

INTERVENTIONS:
Drug: F16IL2 — F16IL2 dose escalation with provisional doses of 10, 20 and 30 Mio IU on Day 1, 8, 15 and 22 of each cycle through a rate-controlled intravenous infusion of 3 hours
Drug: BI 836858 — BI 836858 dose escalation with provisional doses of 10, 20, 40, 80 and 160 mg on days 3, 10, 17 and 24 of each cycle through a rate-controlled intravenous infusion up to 5 hours

SUMMARY:
Phase I, open label, single arm, non-randomized, multicenter, prospective dose escalation study in subjects with acute myeloid leukemia relapse after allogeneic hematopoietic stem cell transplantation (alloHSCT).

DETAILED DESCRIPTION:
The aim of the study is to determine a recommended dose for F16IL2 in combination with BI 836858 in AML relapse after alloHSCT and investigating safety and tolerability of the combination regimen.

Dose escalation will be guided by a Bayesian logistic regression model (BLRM) with overdose control that will be fitted to binary toxicity outcomes. The estimate of parameters will be updated as data are accumulated using the BLRM. At the end of the dose escalation phase, the probability of toxicity at each dose combination level will be calculated to determine an estimate of the MTD. Once the MTD or a biological active dose has been defined, additional patients (up to 10) will be treated with F16IL2 and BI 836858 dosed at this dose combination in order to confirm the safety profile of the combination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with de novo or secondary AML according to the WHO/FAB classification relapsing after alloHSCT, and fulfilling at least one of the following:

   1. bone marrow blasts ≥ 5% of all nucleated cells
   2. appearance of blasts in the peripheral blood
   3. extramedullary AML relapse
2. Age 18 - 75 years.
3. ECOG ≤ 2.
4. Documented negative test for HIV-HBV-HCV. For HBV serology: the determination of HBsAg, anti-HBsAg-Ab and anti-HBCAg-Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV-DNA is required.
5. Negative serum pregnancy test for females of childbearing potential* within 14 days of starting treatment.
6. Informed consent personally signed and dated to participate in the study.
7. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

   * Women of childbearing potential (WOCBP) must be using, from the screening to six months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesteron-only or combined (estrogen- and progesteron-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomized partner or sexual abstinence. Pregnancy test will be repeated at the end of treatment visit.

Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy)

Exclusion Criteria:

1. Known central nervous system manifestation of AML.
2. Previous treatment (e.g., stem cell transplantation, chemotherapy, radiotherapy, investigational drugs) within 4 weeks or a minimum of 5 half-lifes of the treatment, whatever is shorter, of the first study drug intake for this current AML relapse after alloHSCT, except hydroxyurea to control peripheral cell counts up to one day before study medication.
3. Active GvHD requiring systemic immunosuppression, unless controlled with low dose steroids equivalent to a maximum of 10 mg methylprednisolone per day.
4. Chronically impaired renal function (estimated creatinine clearance < 30 ml/min).
5. Inadequate liver function (ALT, AST, ALP or total bilirubin ≥ 3.0 x ULN), if not caused by leukemic infiltration.
6. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
7. History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
8. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
9. Irreversible cardiac arrhythmias requiring permanent medication.
10. Uncontrolled hypertension.
11. Ischemic peripheral vascular disease (Grade IIb-IV).
12. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
13. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of study treatment.
14. Pregnancy or breast-feeding.
15. Requirement of chronic administration of corticosteroids. However, low dose corticosteroids (maximum 10 mg methylprednisolone or equivalent per day when administered for GVHD) are allowed.
16. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
17. Known active or latent tuberculosis (TB).
18. Known hereditary fructose intolerance.
19. Concurrent malignancies other than AML (except basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the patient has been disease-free for at least 2 years.
20. Concomitant treatment with angiogenesis inhibitors or other drugs with proven anti-leukemic activity.
21. Prior treatment with CD33 antibody.
22. Serious, non-healing wound, ulcer or bone fracture.
23. Allergy to study medication or excipients in study medication.
24. Concurrent use of other anti-cancer treatments or agents.
25. Failure to fulfil inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events that are related to treatment and classified as DLTs for each administered dosage | Safety assessment will be performed from day 1 up to day 28 of the Cycle 1 (each cycle is 28 days) for every patient until the end of the enrollment
  To assess the dose limiting toxicity (DLT), maximum tolerated dose (MTD) and recommended dose (RD) of F16IL2 combined with BI 836858

SECONDARY OUTCOMES:
Overall response rate (ORR) | 1) from week 4 up to week 24, every 4 weeks; 2) for EoT: at week 26 (only induction) or 50 (plus maintenance); 3) for follow-up: from week 28 (only induction) or 52 (plus maintenance) up to week 76, every 4 weeks
Relapse-free survival (RFS) | 1) from week 4 up to week 24, every 4 weeks; 2) for EoT: at week 26 (only induction) or 50 (plus maintenance); 3) for follow-up: from week 28 (only induction) or 52 (plus maintenance) up to week 76, every 4 weeks
Time to response (CR or CRi) of responding patients | 1) from week 4 up to week 24, every 4 weeks; 2) for EoT: at week 26 (only induction) or 50 (plus maintenance); 3) for follow-up: from week 28 (only induction) or 52 (plus maintenance) up to week 76, every 4 weeks
Overall survival (OS) rate | From day 1 up to week 76, every 4 weeks
Rate to complete donor chimerism | 1) day 0; 2) from week 4 up to week 24, every 4 weeks; 3) for EoT: at week 26 (only induction) or 50 (plus maintenance); 4) for follow-up: from week 28 (only induction) or 52 (plus maintenance) up to week 76 every 4 weeks
Time to complete donor chimerism | 1) day 0; 2) from week 4 up to week 24, every 4 weeks; 3) for EoT: at week 26 (only induction) or 50 (plus maintenance); 4) for follow-up: from week 28 (only induction) or 52 (plus maintenance) up to week 76 every 4 weeks
Maximum drug concentration [Cmax] | Cycle 1,1) at day 1,2 (week 1); 2) at day 22,23 (week 4)
  Pharmacokinetics assessment of F16IL2 through blood sampling
Time to reach maximum drug concentration [Tmax] | Cycle 1,1) week 1; 2) week 4
  Pharmacokinetics assessment of F16IL2 through blood sampling
Terminal half-life [t1/2] | Cycle 1,1) at day 1,2 (week 1); 2) at day 22,23 (week 4)
  Pharmacokinetics assessment of F16IL2 through blood sampling
Area under the drug concentration-time curve [AUC(0 - t last)] and area under the drug concentration-time curve, extrapolated to infinity [AUC] | Cycle 1, 1) at day 1,2 (week 1); 2) at day 22,23 (week 4)
  Pharmacokinetics assessment of F16IL2 through blood sampling
Accumulation ratio for AUC [R AUC], Cmax [Rmax] and Cmin [R min] | Cycle 1,1) at day 1,2 (week 1); 2) at day 22,23 (week 4)
  Pharmacokinetics assessment of F16IL2 through blood sampling
Total clearance following the dose administered [CL] | Cycle 1,1) at day 1,2 (week 1); 2) at day 22,23 (week 4)
  Pharmacokinetics assessment of F16IL2 through blood sampling
Volume of distribution at steady state [Vss] | Cycle 1,1) at day 1,2 (week 1); 2) at day 22,23 (week 4)
  Pharmacokinetics assessment of F16IL2 through blood sampling
Mean residence time [MRT] | Cycle 1,1) at day 1,2 (week 1); 2) at day 22,23 (week 4)
  Pharmacokinetics assessment of F16IL2 through blood sampling
Maximum drug concentration [Cmax] | Cycle 1 [at day 3,4,6 (week 1); at day 24,25,27 (week 4)]
  Pharmacokinetics assessment of BI 836858 through blood sampling
Time to reach maximum drug concentration [Tmax] | Cycle 1 [at day 3,4,6 (week 1); at day 24,25,27 (week 4)]
  Pharmacokinetics assessment of BI 836858 through blood sampling
Terminal half-life [t1/2] | Cycle 1 [at day 3,4,6 (week 1); at day 24,25,27 (week 4)]
  Pharmacokinetics assessment of BI 836858 through blood sampling
Area under the drug concentration-time curve [AUC(0 - t last)] and area under the drug concentration-time curve, extrapolated to infinity [AUC] | Cycle 1 [at day 3,4,6 (week 1); at day 24,25,27 (week 4)]
  Pharmacokinetics assessment of BI 836858 through blood sampling
Accumulation ratio for AUC [R AUC], Cmax [Rmax] and Cmin [R min] | Cycle 1 [at day 3,4,6 (week 1); at day 24,25,27 (week 4)]
  Pharmacokinetics assessment of BI 836858 through blood sampling
Total clearance following the dose administered [CL] | Cycle 1 [at day 3,4,6 (week 1); at day 24,25,27 (week 4); up to week 21, 22, 23, 24 of Cycle 6, every 4 weeks]
  Pharmacokinetics assessment of BI 836858 through blood sampling
Volume of distribution at steady state [Vss] | Cycle 1 [at day 3,4,6 (week 1); at day 24,25,27 (week 4)]
  Pharmacokinetics assessment of BI 836858 through blood sampling
Mean residence time [MRT] | Cycle 1 [at day 3,4,6 (week 1); at day 24,25,27 (week 4)]
  Pharmacokinetics assessment of BI 836858 through blood sampling
Human anti-fusion protein antibodies (HAFA) levels | 1) at day 1 of every 28 day cycle, from Cycle 1 up to Cycle 12; 2) for EoT: at week 26 (only induction) or 50 (plus maintenance); 3) for follow-up: at week 28 (only induction) or 52 (plus maintenance)
BI 836858 anti-drug antibodies (ADAs) levels | From Cycle 1 to Cycle 6, [at day 3 (week 1); at day 10 (week 2); at day 17 (week 3); at day 24 (week 4)]
The rate of acute and chronic GvHD | From day 1 up to week 76, every 4 weeks
The severity of acute and chronic GvHD | From day 1 up to week 76, every 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Münster University Hospital, Münster